CLINICAL TRIAL: NCT05163067
Title: Combined Aerobic Exercise and Cognitive Training for Alzheimer's Disease Prevention in Seniors With Genetic Susceptibility Estimated by Polygenic Risk Models: Cognition and Neural Plasticity Effects
Brief Title: Combined Aerobic Exercise and Cognitive Training in Seniors With Genetic Susceptibility for Alzheimer's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ICND20210820
Record Dates: First submitted 2021-11-22; First posted 2021-12-20 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2022-11

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; cognitive training; prevention; aerobic exercise; genetic susceptibility; neural plasticity
MeSH Terms: conditions — Alzheimer Disease; Genetic Predisposition to Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined aerobic exercise and cognitive training program (Experimental)
  Interventions: Behavioral: Combined aerobic exercise and cognitive training program
- Standard health counseling at baseline (No Intervention)

INTERVENTIONS:
Behavioral: Combined aerobic exercise and cognitive training program — Participants will take part in a combined aerobic exercise and cognitive training program. The program will include moderate cycling exercise and cognitive game resolving at the same time. The tasks will be instructed and supervised by a fitness expert and a trained clinical neuropsychologist.
  Arms: Combined aerobic exercise and cognitive training program

SUMMARY:
The study aims to investigate the effect of a long-term combined aerobic exercise and cognitive training program on cognitive function, daily function, psychosocial status, and neural plasticity in seniors with genetic susceptibility for Alzheimer's Disease.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is the most common type of dementia and the leading cause of disability in people older than 65 years worldwide. However, there is no effective disease-modifying therapy currently. Therefore, improvement of cognitive function in people at risk and, potentially, prevention of cognitive decline has been gaining attraction.

Our previous research reported a model of a combination single nucleotide polymorphism (SNP) (rs3777215, rs234434, rs71352238, and rs4420638) can predict AD onset with high performance, which is useful to identify people at risk for AD and thus allows for timely treatment and prevention.

Both aerobic exercise and cognitive training have been demonstrated beneficial effects on cognition in subjects with AD and healthy populations. Moreover, the synergistic effects of the combination have been proven recently. However, the effect of combined aerobic exercise and cognitive training on seniors with genetic susceptibility for AD remains to be elucidated. Herein, this study aims to

1. assess the effects of long-term combined aerobic exercise and cognitive training on cognitive function, daily function, psychosocial status, and neural plasticity in seniors with single nucleotide polymorphism of rs3777215, rs234434, rs71352238, and rs4420638.
2. confirm the predictive value of the SNP model for AD in a longitudinal setting.

ELIGIBILITY:
Inclusion Criteria:

* Mandarin-speaking subjects.
* Not clinically demented.
* Meeting the cutoff values of MMSE and CDR.
* With positive variation of rs3777215, rs234434, rs71352238, and rs4420638.

Exclusion Criteria:

* Had major neurologic diagnosis (e.g., Parkinson's disease, stroke, encephalitis, and epilepsy) or other condition that might impair cognition or confound assessments.
* Had a history of psychotic episodes or had major depression (Hamilton Depression Rating Scale score > 24 points).
* Had severe systemic diseases, such as tumors, cardiovascular or orthopedic disorder that can affect the ability to perform the proposed intervention tasks.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2034-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive function over time as assessed by the Montreal Cognitive Assessment (MoCA) | baseline time, year 1, year 3, year 5, year 7
  MoCA will be performed to evaluate the cognition of participants at the enrollment and year 1, year 3, year 5, year 7. The score ranges from 0 to 30, with higher values indicating better cognition.
Change in cognitive function over time as assessed by Mini Mental State Examination (MMSE) | baseline time, year 1, year 3, year 5, year 7
  MMSE will be performed to evaluate the cognition of participants at the enrollment and year 1, year 3, year 5, year 7. The score ranges from 0 to 30, with higher values indicating better cognition.
Change in cognitive function over time as assessed by Clinical Dementia Rating (CDR) | baseline time, year 1, year 3, year 5, year 7
  CDR will be performed to evaluate the cognition of participants at the enrollment and year 1, year 3, year 5, year 7. The score ranges from 0 to 18, with higher values indicating worse cognition.
Change in cognitive function over time as assessed by Verbal Fluency Test | baseline time, year 1, year 3, year 5, year 7
  Verbal Fluency Test will be performed to evaluate the semantic memory function of participants at the enrollment and year 1, year 3, year 5, year 7. Participants are asked to produce as many animals as possible within 1 minute. The score is the number of animals, with higher scores indicating better cognition.
Change in cognitive function over time as assessed by Digit Span Test-Forward and Backward | baseline time, year 1, year 3, year 5, year 7
  Digit Span Tests will be performed to evaluate the working memory of participants at the enrollment and year 1, year 3, year 5, year 7. The total scores are twelve for each test, with higher values indicating better cognition.
Change in cognitive function over time as assessed by Trail-Making Test Parts A and B (TMT-A and TMT-B) | baseline time, year 1, year 3, year 5, year 7
  TMT-A and TMT-B will be performed to evaluate the executive function of participants at the enrollment and year 1, year 3, year 5, year 7. Scoring is based on time taken to complete the test (e.g., 35 seconds yielding a score of 35), with lower scores indicating better cognition.
Change in cognitive function over time as assessed by Boston Naming Test (BNT) | baseline time, year 1, year 3, year 5, year 7
  BNT will be performed to evaluate the language function of participants at the enrollment and year 1, year 3, year 5, year 7. The score ranges from 0 to 30, with higher values indicating better cognition.
Change in cognitive function over time as assessed by California Verbal Learning Test (CVLT) | baseline time, year 1, year 3, year 5, year 7
  CVLT will be performed to evaluate the memory function of participants at the enrollment and year 1, year 3, year 5, year 7. Participants are asked to finish immediate recall, delayed recall, and delayed recognition tasks in the test, with higher scores indicating better cognition.
Change in cognitive function over time as assessed by the Rey-Osterrieth Complex Figure Test (ROCF) | baseline time, year 1, year 3, year 5, year 7
  ROCF will be performed to evaluate the visuospatial function and other cognition domains of participants at the enrollment and year 1, year 3, year 5, year 7. Participants are asked to produce a complicated line drawing, with higher scores indicating better cognition.
The area under curve of the SNP model (rs3777215, rs234434, rs71352238 and rs4420638) for the accurate diagnosis of AD | up to 7 years
  The area under curve is used to show the ability of the SNP model (rs3777215, rs234434, rs71352238 and rs4420638) to diagnose AD. The value of area under curve is higher, then the ability of the SNP model to diagnose AD is stronger.

SECONDARY OUTCOMES:
Change in whole brain volume as accessed by brain MRI | baseline time, year 1, year 3, year 5, year 7
  Brain MRI will be performed to evaluate the whole brain volume of participants at the enrollment and year 1, year 3, year 5, year 7. Whole brain volume is measured in mL and determined by Freesurfer analysis. There is no defined maximum. Zero is the theoretical minimum. Greater number indicates larger brain volume.
Change in daily function over time as assessed by Activities of daily living (ADL) | baseline time, year 1, year 3, year 5, year 7
  ADL will be performed to evaluate the daily function of participants at the enrollment and year 1, year 3, year 5, year 7. The score ranges from 14 to 64, with lower values indicating better function.
Change in anxiety over time as assessed by Hamilton Anxiety Rating Scale (HAMA) | baseline time, year 1, year 3, year 5, year 7
  HAMA will be performed to evaluate the daily function of participants at the enrollment and year 1, year 3, year 5, year 7. The score ranges from 0 to 64, with higher values indicating more severe anxiety.
Change in depression over time as assessed by Hamilton Depression Scale (HAMD) | baseline time, year 1, year 3, year 5, year 7
  HAMD will be performed to evaluate the daily function of participants at the enrollment and year 1, year 3, year 5, year 7. The score ranges from 0 to 96, with higher values indicating more severe depression.
Change in neuropsychiatric symptoms over time as assessed by Neuropsychiatric Inventory Questionnaire (NPI-Q) | baseline time, year 1, year 3, year 5, year 7
  NPI-Q will be performed to evaluate the daily function of participants at the enrollment and year 1, year 3, year 5, year 7. The score ranges from 0 to 144, with higher values indicating more severe neuropsychiatric symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Longfei Jia, MD,PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jia L, Li F, Wei C, Zhu M, Qu Q, Qin W, Tang Y, Shen L, Wang Y, Shen L, Li H, Peng D, Tan L, Luo B, Guo Q, Tang M, Du Y, Zhang J, Zhang J, Lyu J, Li Y, Zhou A, Wang F, Chu C, Song H, Wu L, Zuo X, Han Y, Liang J, Wang Q, Jin H, Wang W, Lu Y, Li F, Zhou Y, Zhang W, Liao Z, Qiu Q, Li Y, Kong C, Li Y, Jiao H, Lu J, Jia J. Prediction of Alzheimer's disease using multi-variants from a Chinese genome-wide association study. Brain. 2021 Apr 12;144(3):924-937. doi: 10.1093/brain/awaa364. PMID 33188687
- [Background] Jia L, Quan M, Fu Y, Zhao T, Li Y, Wei C, Tang Y, Qin Q, Wang F, Qiao Y, Shi S, Wang YJ, Du Y, Zhang J, Zhang J, Luo B, Qu Q, Zhou C, Gauthier S, Jia J; Group for the Project of Dementia Situation in China. Dementia in China: epidemiology, clinical management, and research advances. Lancet Neurol. 2020 Jan;19(1):81-92. doi: 10.1016/S1474-4422(19)30290-X. Epub 2019 Sep 4. PMID 31494009
- [Background] Hill NT, Mowszowski L, Naismith SL, Chadwick VL, Valenzuela M, Lampit A. Computerized Cognitive Training in Older Adults With Mild Cognitive Impairment or Dementia: A Systematic Review and Meta-Analysis. Am J Psychiatry. 2017 Apr 1;174(4):329-340. doi: 10.1176/appi.ajp.2016.16030360. Epub 2016 Nov 14. PMID 27838936
- [Background] Lopez-Ortiz S, Valenzuela PL, Seisdedos MM, Morales JS, Vega T, Castillo-Garcia A, Nistico R, Mercuri NB, Lista S, Lucia A, Santos-Lozano A. Exercise interventions in Alzheimer's disease: A systematic review and meta-analysis of randomized controlled trials. Ageing Res Rev. 2021 Dec;72:101479. doi: 10.1016/j.arr.2021.101479. Epub 2021 Sep 30. PMID 34601135
- [Background] Ben Ayed I, Castor-Guyonvarch N, Amimour S, Naija S, Aouichaoui C, Ben Omor S, Tabka Z, El Massioui F. Acute Exercise and Cognitive Function in Alzheimer's Disease. J Alzheimers Dis. 2021;82(2):749-760. doi: 10.3233/JAD-201317. PMID 34092631